CLINICAL TRIAL: NCT03463135
Title: A Randomized, Multicenter, 3-arm, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacodynamics of Repeated Sublingual Daily Administration of SAR439794 in Peanut Allergic Adult and Adolescent Patients
Brief Title: A Study to Assess Primarily the Tolerability and Safety of SAR439794 After Repeated Sublingual Daily Administration in Peanut Allergic Adult and Adolescent Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDR14287; U1111-1200-1824 (Other: UTN)
Record Dates: First submitted 2018-03-02; First posted 2018-03-13 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — glucopyranosyl lipid-A; gamma-carboxyglutamyl-gamma-carboxyglutamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SAR439794 [PE SLIT + GLA)] (Experimental): GLA repeated doses then SLIT PE escalating doses once daily for 12 weeks
  Interventions: Drug: Glucopyranosyl Lipid A (GLA); Drug: Sublingual Immuno Therapy (SLIT) Peanut Extract (PE)
- Placebo for GLA + SLIT PE (Experimental): Placebo for GLA repeated doses then SLIT PE escalating doses once daily for 12 weeks
  Interventions: Drug: Sublingual Immuno Therapy (SLIT) Peanut Extract (PE); Drug: Placebo for GLA
- Placebo for GLA + Placebo for SLIT PE (Placebo Comparator): Placebo for GLA repeated doses then Placebo for SLIT PE escalating doses once daily for 12 weeks
  Interventions: Drug: Placebo for GLA; Drug: Placebo for SLIT PE

INTERVENTIONS:
Drug: Glucopyranosyl Lipid A (GLA) — Pharmaceutical form:Colloidal aqueous dispersion Route of administration: Sublingual
  Arms: SAR439794 [PE SLIT + GLA)]
Drug: Sublingual Immuno Therapy (SLIT) Peanut Extract (PE) — Pharmaceutical form:Solution Route of administration: Sublingual
  Arms: Placebo for GLA + SLIT PE; SAR439794 [PE SLIT + GLA)]
Drug: Placebo for GLA — Pharmaceutical form:Colloidal aqueous dispersion Route of administration: Sublingual
  Arms: Placebo for GLA + Placebo for SLIT PE; Placebo for GLA + SLIT PE
Drug: Placebo for SLIT PE — Pharmaceutical form:Solution Route of administration: Sublingual
  Arms: Placebo for GLA + Placebo for SLIT PE

SUMMARY:
Primary Objective:

To assess tolerability and safety of SAR439794 [peanut extract (PE) sublingual immunotherapy (SLIT) adjuvanted with Glucopyranosyl Lipid A (GLA)] after repeated sublingual (SL) daily administration in peanut allergic adult and adolescent patients.

Secondary Objective:

To assess pharmacodynamics of SAR439794 after repeated SL daily administration in peanut allergic adult and adolescent patients.

DETAILED DESCRIPTION:
The total study duration per participant is approximately from 15 to 18 weeks (core study) from screening until end-of-study visit, and 2 phone calls at Week 26 and Week 52 after the last Investigational Medicinal Product (IMP) dose.

ELIGIBILITY:
Inclusion criteria :

* Male or female patients, between 18 and 55 years of age, inclusive and adolescents between 12 and 17 years of age (after enrollment of 20 adult patients completed the 6 weeks dose escalation period and the safety and tolerability is deemed acceptable).
* Physician-diagnosed peanut allergy OR convincing history of objective clinical symptoms consistent with immediate hypersensitivity within 4 hours following known ingestion of peanuts or peanut-containing food AND by the following combined criteria:
* Peanut-specific IgE (P-sIgE) >5 kUA/L and Arah2-specific IgE (Arah2-sIgE) >2 kUA/L,
* Skin Prick Test (SPT) to peanut allergen ≥5 mm compared to saline control.
* High-sensitivity C reactive protein (hs-CRP), fibrinogen and neutrophil count within laboratory normal range unless the Investigator considers an abnormality to be clinically irrelevant.
* Ability to perform spirometry based on the American Thoracic Society guidelines.
* Patient must be trained on the proper use of an injectable epinephrine device and should be able to use it.

Exclusion criteria:

* Any history or presence of autoimmune, cardiovascular disease, chronic lung disease, malignancy, psychiatric illness, or gastrointestinal inflammatory conditions, including celiac disease, inflammatory bowel disease and eosinophilic gastrointestinal disorders.
* History of severe anaphylaxis, documented hypotension, neurological compromise (confusion, loss of consciousness), or incontinence known or suspected to be caused by ingestion of peanut or that required treatment with 2 or more administrations of epinephrine or hospitalization.
* Daily oral steroid use for >1 month during the past year, burst oral steroid course in the past 6 months, or >1 burst oral steroid course in the past year.
* Asthma requiring >1 hospitalization in the past year or >1 emergency department visit in the past 6 months.
* Severe or poorly controlled atopic dermatitis.
* Diagnosis of eosinophilic esophagitis.
* Diagnosis of other severe or complicating medical problems.
* Primary immune deficiency.
* If female, pregnancy (defined as positive β-HCG [human chorionic gonadotropin] blood test), breastfeeding.
* If female of childbearing potential, unable to use an effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
* Use of beta blockers, angiotensin converting enzyme inhibitors, angiotensin receptor blockers, or monoamine oxidase inhibitors.
* Any patient who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any patient who cannot be contacted in case of emergency.
* Any patient who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B virus core antibodies (anti-HBc Ab), anti-hepatitis C virus antibodies (anti-HCV Ab), anti-human immunodeficiency Virus 1 and 2 antibodies (anti-HIV1 and anti- HIV2 Ab).
* Presence of sublingual epithelium and oral mucosa wound or infection (abcess, ulcer, candidiasis, gingivitis, etc.) or painful tooth decay.
* Participation in any food immunotherapy interventional study within the past 6 months.
* Patients who had received any monophosphoryl lipid (MPL)- or glucopyranosyl lipid A (GLA)-containing products within the last 6 months.
* Patients who experienced a Grade 3 or higher treatment emergent adverse event following administration of a MPL- or GLA-containing product.
* Use within the past 6 months of systemic immunomodulatory treatment and biologics with an immune target, including Xolair®.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Up to Week 52
  Number of participants with AEs

SECONDARY OUTCOMES:
Assessment of pharmacodynamic (PD) parameter: Peanut-specific serum Immunoglobulin G (IgG) levels | Baseline to Day 85
  Change from baseline to Day 85 in peanut-specific serum IgGs levels in patients administered with Glucopyranosyl Lipid A (GLA) + Sublingual Immuno Therapy Peanut Extract (SLIT PE) versus placebo for GLA + SLIT PE
Assessment of PD parameter: Peanut-specific serum IgG levels | Baseline to Day 57
  Change from baseline to Day 57 in peanut-specific serum IgGs levels (total P-sIgGs, P-sIgG4 and P-sIgG1) in patients administered with GLA + SLIT PE versus placebo for GLA + SLIT PE
Assessment of PD parameter: Peanut-specific serum Immunoglobulin E (IgE) levels | Baseline to Day 57, Baseline to Day 85
  Change from baseline to Day 57 and Day 85 in peanut-specific IgE in patients administered with GLA + SLIT PE versus placebo for GLA + SLIT PE
Assessment of PD parameter: Skin Prick Test | On Day 85
  Absolute change from baseline in Skin Prick Test (SPT) to peanut allergen at Day 85 only in patients administered with GLA + SLIT PE versus placebo for GLA + SLIT PE
Maximum SLIT PE dose | On Day 85
  Maximum SLIT PE dose reached by patients administered with GLA + SLIT PE versus placebo GLA + SLIT PE

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (16):
  - Investigational Site Number 8400004, Little Rock, Arkansas
  - Investigational Site Number 8400019, Mission Viejo, California
  - Investigational Site Number 8400008, San Diego, California
  - Investigational Site Number 8400020, San Jose, California
  - Investigational Site Number 8400006, Stanford, California
  - Investigational Site Number 8400013, Denver, Colorado
  - Investigational Site Number 8400014, Louisville, Kentucky
  - Investigational Site Number 8400002, Baltimore, Maryland
  - Investigational Site Number 8400001, Boston, Massachusetts
  - Investigational Site Number 8400009, Minneapolis, Minnesota
  - Investigational Site Number 8400016, Minneapolis, Minnesota
  - Investigational Site Number 8400010, Charleston, North Carolina
  - Investigational Site Number 8400011, Cincinnati, Ohio
  - Investigational Site Number 8400012, Medford, Oregon
  - Investigational Site Number 8400003, Seattle, Washington
  - Investigational Site Number 8400017, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org